CLINICAL TRIAL: NCT04358146
Title: Study on the Efficacy and Tolerance of a New Anti-regurgitation Infant Formula: a Double-blind, Randomized, Controlled, International, Multi-centric Clinical Trial
Brief Title: Study on the Efficacy and Tolerance of a New Anti-regurgitation Infant Formula (STELLAR)
Acronym: STELLAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: United Pharmaceuticals (Industry)
Collaborators: Statitec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UP2017-04-STELLAR
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Gastroesophageal Reflux in Children
Keywords: Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — locust bean gum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): new thickened infant formula containing fibres
  Interventions: Other: Experimental Infant formula
- Control (Active Comparator): infant formula thickened with locust bean
  Interventions: Other: Infant formula thickened with locust bean gum

INTERVENTIONS:
Other: Experimental Infant formula — Exclusive formula feeding with the new infant formula thickened with fibers
  Arms: Test
Other: Infant formula thickened with locust bean gum — Exclusive formula feeding with the formula thickened with locust bean
  Arms: Control

SUMMARY:
The aim of the study is to assess the effectiveness of this new formula on regurgitations and secondarily its effect on digestive tolerance through a randomized, controlled, double-blind trial against a comparator.

DETAILED DESCRIPTION:
The study duration is 1 month and 2 days. It is possible to add 2 additional months (optional).

The 2 first days (from D-3 to D0) correspond to the pre-selection period. These 2 days are followed by the follow-up month (from D0 to D30). It is possible to add an optional follow up of 2 months (form D30 to D90).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 2 regurgitation episodes per day during the last 2 weeks and ≥ 4 regurgitation episodes per day in average during the last 2 days,
* exclusive or predominant formula feeding
* whose parents signed informed consent

Exclusion Criteria:

* preterm infants or birthweight <2500g
* Post enteritis lactose intolerance
* Suspected or diagnosed cow's milk protein allergy requiring an eviction diet
* Use of medications that may interfere with regurgitation or gastrointestinal transit (such as alginates, laxatives, antibiotics...). All these medications have to be stopped at least 7 days before inclusion visit (V1)
* Infants presenting with any situation which, according to the investigator, may interfere with the study participation, or lead to a particular risk for the subject

Ages: 2 Weeks to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 346 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of regurgitation | Day 14
  Decrease of the daily number of regurgitation between baseline and day 14

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papadopoulou, Study Director — University of Athens, Athens Children's Hospital "AGIA SOFIA"